CLINICAL TRIAL: NCT01331551
Title: Crossover Study on Human Exposure to Phthalates and Male Fertility
Brief Title: Mesalamine and Reproductive Health Study
Acronym: MARS
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Boston Children's Hospital (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Russ Hauser, Principal Investigator, Harvard School of Public Health (HSPH)
Other Study IDs: 5R01ES17285-2; 5R01ES017285 (NIH)
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Colitis Ulcerative; Crohn Disease
Keywords: Inflammatory Bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for hormones, urine for phthalates, semen for DNA and RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- men with inflammatory bowel disease: Men between the ages of 18-55 with inflammatory bowel disease who are taking mesalamine medication.

SUMMARY:
The purpose of this study is to investigate the relationship of high exposure to dibutyl phthalate (DBP) from the use of Asacol with clinical and intermediate markers of male fertility, including semen quality, sperm DNA damage, transcript profiles of sperm mRNA and sncRNAs, and reproductive hormones.

Hypothesis 1: High exposure to DBP from the use of Asacol is associated with decreased sperm concentration and motility, and increased sperm DNA damage.

Hypothesis 2: High exposure to DBP from the use of Asacol is associated with decreased serum testosterone, altered LH:testosterone ratio, and decreased inhibin-B.

Hypothesis 3: High exposure to DBP from the use of Asacol is associated with altered transcript profiles of sperm mRNAs and sncRNAs.

DETAILED DESCRIPTION:
There are 2 ways you can participate in the study.

OPTION 1 involves 6 one-hour visits to the Massachusetts General Hospital (MGH) Andrology Clinic over a 9 month period. At each visit you would be asked to fill out questionnaires and to provide a urine, semen, and blood sample. Following Visit 2, you are asked to switch your brand of mesalamine medication. After 4 months, you change back to your original brand of medication. The change in medication will be done in consultation with your primary GI doctor. If the cost of co-payment is greater for the new brand of medication, we will provide compensation to cover the difference. In the case you do not have prescription drug health insurance coverage, the study will reimburse up to $4000 to cover the cost for Asacol, Pentasa or Lialda medication taken during your study participation.

OPTION 2 involves 4 one-hour visits to MGH Andrology clinic. At each visit you complete questionnaires and provide a blood, urine and semen sample. You are eligible for Option 2 if you are currently taking Asacol or Asacol HD and do not want to change your medication.

ELIGIBILITY:
Inclusion Criteria:

* Must be taking mesalamine medication. Willing to switch brand of medication for 4 months or currently taking Asacol or Asacol HD.
* Has not taken steroid medication within the previous 3 months. Is able to come to MGH hospital for 6 visits.

Exclusion Criteria:

* Is not taking mesalamine medication. Unwilling to switch brand of medication for 4 months.
* Is or has taken steroid medication within the past 3 months. Is unable to come to MGH hospital for 6 visits.
* Has had a vasectomy or has documented infertility.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Men between the ages of 18-55 who have inflammatory bowel disease.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Altered semen quality and sperm transcriptome analysis | Initial analysis takes place approximately 4-5 months after patient enrolls and after he has completed first crossover of medication. The second phase takes place about 8-10 months later after he crosses back to original medication.

SECONDARY OUTCOMES:
Serum levels of reproductive hormones | Analysis of hormone levels take place at the same intervals described above, 4-5 months after enrollment and then again 8-10 months after enrollment when patient has resumed taking orginal medication.

CONTACTS AND LOCATIONS:
Overall Officials: Russ B Hauser, MD, ScD, MPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Massachuetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants may receive semen and hormone analysis if they desire.